CLINICAL TRIAL: NCT04368247
Title: Skin Fluorescent Imaging (SFI) System in Patients With Nevi
Status: Completed | Type: Observational
Sponsor: Orlucent, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SFI 003
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Nevus; Dysplasia; Epithelial
Keywords: Nevus; Atypical Nevi; Mole; Skin Imaging
MeSH Terms: conditions — Nevus; Carcinoma in Situ; Dysplastic Nevus Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — If the Site specific pathology lab will not allow the sponsor to make a digital image of the original slide, then the Sponsor is asking that a duplicate slide be provided for digital scanning. Once scanning is complete these additional slides may not be returned to the site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Nevi undergoing biopsy per SOC: Subjects with Nevi who will as part of their standard of care, will undergo biopsy.
  Interventions: Diagnostic Test: Skin Fluorescent Imaging

INTERVENTIONS:
Diagnostic Test: Skin Fluorescent Imaging — Application of reagents, then imaging and scoring
  Other Names: SFI 003 Imaging

SUMMARY:
The Sponsor has developed the Skin Fluorescent Imaging (SFI) system, an in vivo imaging modality, for the purpose of providing physicians with insight into the biological changes occurring during tissue remodeling in a nevus.

DETAILED DESCRIPTION:
The SFI system, a non-invasive point-of-care imaging system, is able to detect markers associated with tissue remodeling and thus provide real-time information about biological and structural changes occurring in nevi indicative of dysplastic transition.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study a subject must meet all of the following criteria:

* Provide a signed and dated informed consent form
* Age ≥ 18 years old
* Subjects must present with suspicious atypical nevi scheduled for a biopsy*
* Nevi with at least 1 cm of skin surrounding the mole
* Nevi must be accessible to the SFI imaging device
* Excisional or a tangential excision with a dept of 1 to 2 mm biopsy will be performed for the mole tested within 21 days of testing.
* Nevi with clinically atypical features

Only 1 mole per eligible subject will be SFI tested in this study. *NOTE: a subset of patients (~10%) with benign nevi (by clinical observation) who wish to have nevi removed for cosmetic reasons will be enrolled as negative controls.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Subjects who are younger than 18 years old
* Lesions that are consistent with

  - Features of Keratosis and keratin plugs
  * Basal Cell Carcinoma
  * Squamous Cell Carcinoma
  * Challenging anatomical location (e.g., body cervices)
* Subjects with nevi that fit the inclusion criteria but are:

  * Less than 1 cm from the eyes
  * On the palms of the hands or soles of the feet
  * Associated with scar tissue
  * Mucosal lesions
  * Ulcerated lesions / breached skin
  * Lesions with some clinical certainty of being melanomas (large, dark, etc.)
  * Any nevi with ink marking including tattoos, on or adjacent to the nevi
  * Lesions treated with local anesthesia such as lidocaine prior to enrollment
  * Lesions larger than 20 mm or too large to allow imaging
  * Subject is known to be pregnant
  * Subject who is mentally or physically unable to comply with all aspects of the study
  * Subject who is undergoing systemic cancer treatment within 6 months of SFI testing
  * Subject with hypersensitivity to any of the SFI reagents
  * Subjects with known sensitivity to fluorescent dyes
  * Any subject who has previously participated (testing to biopsy) in SFI 003

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who present with suspicious nevus/nevi and who require a Standard of Care (SOC) biopsy of the atypical nevi will be able to participate in the study.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Establish the performance of SFI | 1year
  Establish the performance (sensitivity and specificity) for SFI in comparison to dysplasia.

SECONDARY OUTCOMES:
To compare SFI to clinical diagnosis. | 1 year
  Comparison of the SFI score ( 0 to 10) to the clinical diagnosis of the physician assessing and the pathologist
To establish the tolerability of SFI Testing by documenting minimal, transient events that occur with reagent application. | 1 year
  Adverse events will be collected to ensure overall safety of reagents and imaging

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Shachaf, PhD, Study Director — President
Locations (4):
- United States (4):
  - Center for Dermatology Clinical Research, Inc, Fremont, California
  - Quest Dermatology Research, Northridge, California
  - Solano Dermatology Associates, Vallejo, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided